CLINICAL TRIAL: NCT01208519
Title: Impact of Specific Antibiotic Therapies on the Prevalence of Human Host Resistant Bacteria in Hospitalised Patients (SATURN 04)
Brief Title: SATURN 04 Nosocomial Acquisition Study
Acronym: SATURN
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Collaborators: Clinical Centre of Serbia (Other); National Institute of Infectious Diseases Matei Bals (Unknown); University Hospital, Geneva (Other); Canisius-Wilhelmina Hospital (Other); Universiteit Antwerpen (Other)
Responsible Party: Dr. Evelina Tacconelli, Catholic University of the Sacred Heart; Policlinico A. Gemelli, Rome
Other Study IDs: FP7-N° 241796
Record Dates: First submitted 2010-09-23; First posted 2010-09-24 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2012-11

CONDITIONS: Bacterial Resistance; Infection Resistant to Multiple Drugs; Staph Aureus Methicillin Resistant Colonization; Infection Due to ESBL Bacteria
Keywords: Drug resistance, Microbial; Methicillin-Resistant Staphylococcus aureus; ESBL; Colonisation; Screening; Gram-negative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Nasal and rectal swabs
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Case Control Study 1: To define the impact of antibiotics on new acquisition of MRSA and ESBL-producing gram negative bacteria, a matched case-control study will be done (ratio 1:4). The control group will be selected among patients not receiving antibiotics, admitted in the same ward on the day of the corresponding case, with negative cultures at hospital admission. Matching criteria will include: age (±5 years), sex, and total length of hospitalization.
- Case control study 2: To define individual level of risk related to specific antibiotics, patients acquiring MRSA and ESBL-producing gram negative bacteria will be compared with patients not acquiring antibiotic-resistant strains after starting antibiotic therapy (ratio 1:4). Previously known risk factors or clinically relevant significant variables from the univariate analysis will be considered for inclusion in multivariate logistic regression analysis.

SUMMARY:
The study is the WP4 of the EU-funded (7th FW) project SATURN (Impact of Specific Antibiotic Therapies on the prevalence of hUman host ResistaNt bacteria). A total of 6 surgical and 6 medical wards will participate in the study. Sites of the study are located in 3 countries (Italy, Serbia, Romania). This WP will compare nosocomial acquisition rates of methicillin-resistant Staphylococcus aureus (MRSA) and extended-spectrum beta-lactamase (ESBL)-producing gram-negative bacteria (E.coli, Klebsiella spp. and Proteus spp.) among different treatment groups and define the temporal relationship between the start of antibiotic therapy, the acquisition of new colonisation in patients previously not colonised, and the development of a bacterial infection caused by the same strain isolated in a screening sample. This goal will be achieved by completing the following primary objectives:

* To determine the rate of acquisition of target antibiotic-resistant bacteria by 1,000 antibiotic-days according to different classes of antibiotics, duration of therapy and antibiotic combination (monotherapy versus combination therapy);
* To determine genotypic relation between colonising and infecting strain in the same patient and patients' and hospital staff colonising strains (to be performed in collaboration with WP1 of the SATURN project);
* To study the virulence and fitness of the isolates (i.e. new colonising strains) causing subsequent nosocomial infections (to be performed in collaboration with WP1 of SATURN project);
* To predict the risk for nosocomial infections due to target bacteria after a single treatment therapy adjusted by length of hospitalisation and ward colonisation pressure.

DETAILED DESCRIPTION:
Nasal samples for the detection of MRSA and rectal samples (stoma sample in case of colostomy) for ESBL producing gram negative bacteria will be obtained at hospital admission and discharge. Patients starting antibiotic therapy per os and/or intravenously will be sampled at antibiotic start (t0, within one hour) and at the following intervals: day 3 (t1), 7 (t2), 15 (t3), 30 (t4). Patients colonized with MRSA and/or ESBL-producing gram negative bacteria before starting antibiotic therapy (t0 sample) will be excluded from follow-up cultures and analysis. All patients included in the study will be followed to determine whether they develop clinical infections with the target ARB. Patients will be followed during the hospitalization and afterwards for a total of 30-day from the inclusion in the study. Screening will be performed in outpatient clinics after patients' discharge from the hospital within 30 days of starting antibiotic (t0 sample).

Nasal and rectal cultures will be also obtained from the ward staff at the beginning and at the end of the study. This group includes nurses and all staff including doctors having contacts with patients. These cultures will be handled in the same manner as the patients' cultures

ELIGIBILITY:
Inclusion Criteria:

* All hospitalized non ICU patients at hospital admission/discharge;
* Age >18 years old;
* All patients starting intravenous and/or oral antibiotic treatments during hospitalization.

Exclusion Criteria:

* Pregnancy;
* Recent nose surgery (for nasal swabs).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients will be screened at hospital admission and hospital discharge during the study period. Patients colonised with MRSA and/or ESBL-producing gram-negative bacteria before starting antibiotic therapy will be excluded from follow-up cultures and analysis.
  Patients starting antibiotic therapy per os and/or intravenously will be sampled at antibiotic start (t0, within one hour) and at the following intervals: day 3 (t1), 7 (t2), 15 (t3), 30 (t4). Screening will be performed in outpatient clinics after patients' discharge from the hospital.
Sampling Method: Non-Probability Sample
Enrollment: 16680 (Estimated)
Dates: Start 2010-11; Primary Completion 2012-11 (Actual); Study Completion 2015-01

PRIMARY OUTCOMES:
Impact of different antibiotics in selecting antimicrobial resistance in in-patients | 5 years (January 2015)
  Rate of acquisition of target antibiotic-resistant bacteria by 1,000 antibiotic-days in hospitalized patients will be calculated. The rate will be also defined according to antibiotic class and single drug.

SECONDARY OUTCOMES:
Colonization and infection risk according to antibiotic treatment duration | 5 years (January 2015)
  Rate of nosocomial infections by 1,000 days of hospitalization in patients undergoing antibiotic therapy will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Evelina Tacconelli, MD PhD, Study Chair — Università Cattolica del Sacro Cuore - Policlinico A. Gemelli - Roma
Locations (3):
- Università Cattolica del Sacro Cuore; Policlinico A. Gemelli, Rome, Lazio, Italy
- Institute of Infectious Diseases Matei Bals, Bucharest, Romania
- Clinical Center of Serbia, Belgrade, Serbia

REFERENCES:
- [Derived] Niehus R, van Kleef E, Mo Y, Turlej-Rogacka A, Lammens C, Carmeli Y, Goossens H, Tacconelli E, Carevic B, Preotescu L, Malhotra-Kumar S, Cooper BS. Quantifying antibiotic impact on within-patient dynamics of extended-spectrum beta-lactamase resistance. Elife. 2020 May 7;9:e49206. doi: 10.7554/eLife.49206. PMID 32379042
- [Derived] Tacconelli E, Gorska A, De Angelis G, Lammens C, Restuccia G, Schrenzel J, Huson DH, Carevic B, Preotescu L, Carmeli Y, Kazma M, Spanu T, Carrara E, Malhotra-Kumar S, Gladstone BP. Estimating the association between antibiotic exposure and colonization with extended-spectrum beta-lactamase-producing Gram-negative bacteria using machine learning methods: a multicentre, prospective cohort study. Clin Microbiol Infect. 2020 Jan;26(1):87-94. doi: 10.1016/j.cmi.2019.05.013. Epub 2019 May 23. PMID 31128285
- [Derived] Meletiadis J, Turlej-Rogacka A, Lerner A, Adler A, Tacconelli E, Mouton JW; the SATURN Diagnostic Study Group. Amplification of Antimicrobial Resistance in Gut Flora of Patients Treated with Ceftriaxone. Antimicrob Agents Chemother. 2017 Oct 24;61(11):e00473-17. doi: 10.1128/AAC.00473-17. Print 2017 Nov. PMID 28807914
- [Derived] De Angelis G, Restuccia G, Venturiello S, Cauda R, Malhotra-Kumar S, Goossens H, Schrenzel J, Tacconelli E. Nosocomial acquisition of methicillin-resistant Staphyloccocus aureus (MRSA) and extended-spectrum beta-lactamase (ESBL) Enterobacteriaceae in hospitalised patients: a prospective multicenter study. BMC Infect Dis. 2012 Mar 29;12:74. doi: 10.1186/1471-2334-12-74. PMID 22458427
- See also: European Commission website — http://ec.europa.eu/research/health/infectious-diseases/antimicrobial-drug-resistance/projects/014_en.html
- See also: Website of Policlinico A. Gemelli, Roma — http://www.policlinicogemelli.it
- See also: Università Cattolica Sacro Cuore, Roma — http://roma.unicatt.it